CLINICAL TRIAL: NCT04578743
Title: Exercise as Concussion Therapy Trial
Brief Title: Exercise as Concussion Therapy Trial- 2
Acronym: ExACTT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-induced lockdowns.
Sponsor: ANSwers Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ExACTT-2
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Mild Traumatic Brain Injury; Concussion, Mild
Keywords: Concussion; Mild Traumatic Brain Injury (mTBI); Exercise Therapy; Telemedicine; Therapeutic Intervention; Autonomic Function; Medical Device
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: This study is a Phase 2, open-label study of a therapeutic intervention (graded exercise) compared to a reference therapy (passive stretching) in patients who have sustained mTBI. Subjects will be randomly assigned with a ratio of 1:1 to complete either graded exercise or passive stretching using a parallel-group design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Graded Exercise (Experimental): ClearPlay(TM): a novel therapeutic intervention, downloadable to an Apple i-touch or i-phone device, will provide a telemetry-based graded exercise program for 20 minutes each day, identifying a heart rate target that will be advanced weekly for up to 8 weeks as symptoms resolve.
  Interventions: Device: Graded Exercise Therapy: ClearPlay(TM)
- Passive Stretching (Experimental): ClearPlay(TM): we have created a passive stretching program (placebo arm) downloadable to an Apple i-touch or i-phone device, that will provide a telemetry-based guided passive stretching program for 20 minutes each day for up to 8 weeks as symptoms resolve.
  Interventions: Device: Graded Exercise Therapy: ClearPlay(TM)

INTERVENTIONS:
Device: Graded Exercise Therapy: ClearPlay(TM) — ClearPlayTM; a novel therapeutic intervention, downloadable to an Apple i-touch or i-phone device, that provides a telemetry-based graded exercise program that enables remote monitoring of symptoms.

SUMMARY:
This study is a Phase 2, open-label study of a therapeutic intervention (graded exercise)compared to a reference therapy (passive stretching) in patients who have sustained mTBI. Subjects will be randomly assigned with a ratio of 1:1 to complete either graded exercise or passive stretching using a parallel-group design.

The effects of graded exercise and passive stretching will be compared using ClearPlay© (ANSwers Neuroscience Pty Ltd commercial mobile application)

The study will also validate the performance of two devices:

1. ClearHeart©, ANSwers Neuroscience Pty Ltd commercial prototype for cold pressor testing, compared to ice bucket testing.
2. ClearPlay©, ANSwers Neuroscience Pty Ltd commercial prototype based on the joint position error test to assess "whiplash".

DETAILED DESCRIPTION:
Study Type: Interventional Estimated Enrollment: 400 participants Allocation: Randomized Intervention Model: Parallel Assignment Masking: None (Open Label) Primary Purpose: Treatment Official Title: A Therapeutic Intervention, Open-Label Study to Compare the Efficacy and Safety of Graded Exercise Compared to Passive Stretching in Subjects Who Have Sustained a Mild Traumatic Brain Injury Estimated Study Start Date: October 1, 2020 Estimated Primary Completion Date: September 30, 2022 Estimated Study Completion Date: September 30, 2023

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥14 to ≤45, able and willing to provide informed consent (≥18 years), or informed consent is obtained by the parent or legal guardian for minor subjects, with the minor providing age appropriate assent, according to local law and regulations;
2. Subject is fluent in English, able to understand and agree to comply with protocol requirements, and complete all assessments;
3. Subject has a history of recent concussion as diagnosed by a health care professional within 3 to 14 days of enrolment; Note: Concussion is defined as a head injury/blow to the head resulting in any of the following 3 signs and/or new symptoms: (1) amnesia for less than 24 hours; (2) Loss of consciousness for less than 30 minutes; (3) Glasgow Coma Scale score > = 13; (4) Dazed and Confused/bell rung; with at least 1 new symptom or augmentation of a previous symptom on the PCSS as compared with baseline at the time of enrolment, including: headaches, dizziness, fatigue, irritability, insomnia, difficulty concentrating, and/or memory difficulties; (5) The composite symptom score on the PCSS must be at least 3 points higher post-concussion than pre-concussion.
4. Subject has daily access to the internet.

Exclusion Criteria:

1. History of prior head injury as defined by:

   1. An injury/blow to the head within 12 months prior to screening with any associated residual symptoms;
   2. An injury/blow to the head within 3 months prior to screening diagnosed as a concussion;
   3. An injury/blow to the head within 3 months prior to screening with any of the following symptoms: amnesia, loss of consciousness, dazed and confused/bell rung;
2. Evidence of blood or micro-hemorrhages on prior or current computed tomography scan or magnetic resonance imaging scan if obtained;
3. Diagnosis of a neurological condition including the following: stroke, multiple sclerosis, epilepsy, brain tumor/cancer, encephalitis, dementia, movement disorder, or spontaneous nystagmus;
4. Psychiatric history with any of the following:

   1. History of psychiatric hospitalization, history of legal trouble for violence;
   2. Requires psychotropic medication other than (1) stable dose of a selective serotonin reuptake inhibitors (SSRI) medication, or (2) stable dose of a tricyclic antidepressants (TCA) medication;
   3. Prior diagnosis of psychotic disorder, bipolar disorder, eating disorder, substance abuse disorder;
5. Current use of a beta blocker;
6. History of drug or alcohol dependency or abuse within a year before Screening, by self-report;
7. Two or more the following cardiovascular risk factors:

   1. Prior diagnosis of, or currently taking medication for cardiovascular, metabolic or pulmonary conditions;
   2. Family history of myocardial infarction, coronary revascularization or sudden death before 55 years;
   3. Diagnosis of hypertension;
   4. Diagnosis of hyperlipidemia;
   5. Subjects with peripheral circulatory disorders;
8. Subjects who are unable or unwilling to exercise for health or personal reasons;
9. Subjects who have musculoskeletal injuries which could make exercise difficult or painful.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
ExACTT | 2 Years
  The primary objective of the study is to compare the effects of graded exercise and passive stretching using ClearPlayTM (ANSwers Neuroscience Pty Ltd commercial mobile application) on recovery following mTBI in the Australian setting.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Master, MD, Study Director — Children's Hospital of Philadelphia
Locations (3):
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - University of Queensland, Brisbane, Queensland
  - Alfred Health, Melbourne, Victoria

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT04578743/Prot_ICF_000.pdf